CLINICAL TRIAL: NCT05582083
Title: Managed Access Program for Momelotinib in Patients With a Diagnosis of Intermediate or High-risk Myelofibrosis (MF), Including Primary Myelofibrosis (PMF) or Secondary Myelofibrosis (Post- Polycythemia Vera/ Essential Thrombocytopenia (PV/ET)), With Anaemia
Brief Title: Managed Access Program for Momelotinib in Myelofibrosis
Status: No longer available | Type: Expanded Access
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 219595
Record Dates: First submitted 2022-10-12; First posted 2022-10-17 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Myelofibrosis; Primary Myelofibrosis
Keywords: Momelotinib; GSK3070785
MeSH Terms: conditions — Primary Myelofibrosis | interventions — N-(cyanomethyl)-4-(2-((4-(4-morpholinyl)phenyl)amino)-4-pyrimidinyl)benzamide

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Momelotinib — Momelitinib available as tablets.
  Other Names: GSK3070785

SUMMARY:
Compassionate use access to Momelotinib/GSK3070785 for eligible participant with diagnosis of intermediate or high-risk myelofibrosis (MF), including primary myelofibrosis (PMF) or secondary myelofibrosis (post- polycythemia vera/ essential thrombocytopenia (PV/ET)), with anemia.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent can be obtained from the patient or legally authorised representative as per local regulations
* Diagnosis of intermediate or high-risk myelofibrosis (MF), including primary myelofibrosis (PMF) or secondary myelofibrosis (post- polycythemia vera/ essential thrombocytopenia (PV/ET)), with anemia
* 18 years or older (at the time consent is obtained)
* The patient is willing to abide by the contraception requirements.
* No known hypersensitivity to momelotinib, its metabolites, or any of the formulation excipients

Exclusion Criteria:

* Pregnant or breastfeeding female

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline